CLINICAL TRIAL: NCT04189640
Title: The Efficacy of Different Volumes for Ultrasound-Guided Adductor Canal Block for Postoperative Analgesia Management After Total Knee Arthroplasty Surgery
Brief Title: Ultrasound-Guided Adductor Canal Block for Total Knee Arthroplasty Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Medipol Hospital 7
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Knee Osteoarthritis; Knee Arthropathy; Knee Pain Chronic; Knee Deformity; Knee Disease
Keywords: Adductor canal block; Postoperative pain management; Knee arthroplasty surgery
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: There are three models for this study. The first group is 20 ml volume group, the second one is 30 ml group, the third one is 40 ml group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the patient, the investigators and the pain nurse who performs postoperative pain evaluation will blind to the data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 20 = 20 ml volume adductor canal block (Active Comparator): ACB will be performed at the end of the surgery, before extubation. After identifying the adductor canal, by using the in-plane technique, the probe will be placed at the mid-thigh, half the distance between the inguinal crease and the patella, for block location. The superficial femoral artery will be visualized dorsal to the sartorius muscle. Then, the probe will be removed to distally. At this level, the hyperechoic view of the saphenous nerve will be visualized lateral and anterior to the artery in the subsartorial region. 5 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 20ml will be injected here.
  Interventions: Drug: Postoperative analgesia management
- Group 30 = 30 ml volume adductor canal block (Active Comparator): ACB will be performed at the end of the surgery, before extubation. After identifying the adductor canal, by using the in-plane technique, the probe will be placed at the mid-thigh, half the distance between the inguinal crease and the patella, for block location. The superficial femoral artery will be visualized dorsal to the sartorius muscle. Then, the probe will be removed to distally. At this level, the hyperechoic view of the saphenous nerve will be visualized lateral and anterior to the artery in the subsartorial region. 5 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 30ml will be injected here.
  Interventions: Drug: Postoperative analgesia management
- Group 40 = 40 ml volume adductor canal block (Active Comparator): ACB will be performed at the end of the surgery, before extubation. After identifying the adductor canal, by using the in-plane technique, the probe will be placed at the mid-thigh, half the distance between the inguinal crease and the patella, for block location. The superficial femoral artery will be visualized dorsal to the sartorius muscle. Then, the probe will be removed to distally. At this level, the hyperechoic view of the saphenous nerve will be visualized lateral and anterior to the artery in the subsartorial region. 5 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 40ml will be injected here.
  Interventions: Drug: Postoperative analgesia management

INTERVENTIONS:
Drug: Postoperative analgesia management — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure. If the VAS score will be ≥ 4, 0.5 mg/ kg tramadol IV will be administered.

SUMMARY:
The ultrasound-guided selective blockade of the saphenous nerve in the adductor canal provides effective analgesia and reduces postoperative pain in patients undergoing arthroscopic medial meniscectomy. Selective blockade of the saphenous nerve in the adductor canal provides effective analgesia without quadriceps muscle weakness. It has been shown that the adductor canal block (ACB) block increases the spread of local anesthetics in a distal and proximal way. Therefore, the proximal spread of local anesthetics may cause possible quadriceps weakness. The distal spread of local anesthetics may increase analgesic effect via sciatic nerve. The different volumes for ACB is a topic of discussion. The aim of this study is to compare the different volumes of US-guided ACB performing for postoperative analgesia management after total knee arthroplasty surgery.

DETAILED DESCRIPTION:
Knee arthroplasty is one of the most common orthopedic procedures. Patients may complain severe pain due to the surgical trauma and the prosthesis. Opioid agents are commonly used for analgesia management. However, opioids have adverse effects such as nausea, vomiting, sedation and respiratory depression. Peripheral nerve blocks such as femoral block, adductor canal block (ACB) may be performed to reduce opioid consumption and opioid-related side effects.

Selective blockade of the saphenous nerve in the adductor canal for knee surgery provides effective analgesia without quadriceps muscle weakness. This is an important advantage of ACB since it there is no motor blockade in the postoperative period. Blocking of the motor branches leads to delaying of the mobilization and it increases the patient's falling risk. ACB, targets the saphenous nerve and the vastus medialis branch which are the two largest sensorial nerves of the femoral nerve that innervates the knee. ACB blocks the articular branches of the obturator nerve at the same time. Since the ACB is performed at the distal site of thigh it does not target majority of the efferent branches of the quadriceps muscle, therefore the strength of this muscle may not be affected. ACB is usually performed with a volume of 10-30 ml and studies may be needed including different volumes to understand its effectiveness.

The aim of this study is to compare the different volumes (20 ml, 30 ml, and 40 ml) of US-guided ACB for postoperative analgesia management after total knee arthroplasty. The primary aim is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), motor blockage, the first mobilization time, and adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for total knee arthroplasty under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | Change from baseline opioid consumption at postoperative 1, 2, 4, 8, 16, 24 and 48 hours
  The primary aim is to compare perioperative and postoperative opioid consumption

SECONDARY OUTCOMES:
Visual analogue scores (VAS) | Postoperative 1, 2, 4, 8, 16, 24, and 48 hours
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 1, 2, 4, 8, 16, 24 and 48 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not share IPD

REFERENCES:
- [Background] Jiang X, Wang QQ, Wu CA, Tian W. Analgesic Efficacy of Adductor Canal Block in Total Knee Arthroplasty: A Meta-analysis and Systematic Review. Orthop Surg. 2016 Aug;8(3):294-300. doi: 10.1111/os.12268. PMID 27627711
- [Background] Kapoor R, Adhikary SD, Siefring C, McQuillan PM. The saphenous nerve and its relationship to the nerve to the vastus medialis in and around the adductor canal: an anatomical study. Acta Anaesthesiol Scand. 2012 Mar;56(3):365-7. doi: 10.1111/j.1399-6576.2011.02645.x. PMID 22335278
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251